CLINICAL TRIAL: NCT03833791
Title: Effect of the Prescription of Physical Activity on the Fat, Muscle Mass, and Body Weight of Overweight or Adult Men and Women: Randomized Clinical Trial of 6 Month Duration.
Brief Title: Effect of Different Physical Programs on the Body Composition of Adult Men and Women With an Initial Body Fat >25% and >30%, Respectively.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Alberto Hernández de los Reyes, Principal Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TESIS-OBESITICS-2018
Record Dates: First submitted 2019-02-01; First posted 2019-02-07 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Overweight; Obesity
Keywords: obesity; Physical Activity; fat mass; fat free mass
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CON) (Active Comparator): education and modifying diet
  Interventions: Behavioral: education and modifying diet
- Moderate physical activity Group (PAM) (Experimental): education, modifying diet and physical activity prescription
  Interventions: Behavioral: education, modifying diet and physical activity prescription
- Intensity physical activity Group (PAI) (Experimental): education, modifying diet and physical activity prescription
  Interventions: Behavioral: education, modifying diet and physical activity prescription

INTERVENTIONS:
Behavioral: education and modifying diet — The control group maintains a sedentary lifestyle and is only subjected to follow a hypocaloric diet
  Arms: Control Group (CON)
Behavioral: education, modifying diet and physical activity prescription — One group, in addition to fulfilling a hypocaloric diet identical to the control group, is subjected to prescribe moderate physical activity.
  Other group, in addition to fulfilling a hypocaloric diet identical to the control and moderate group, is subjected to prescribe intense activity.
  Arms: Intensity physical activity Group (PAI); Moderate physical activity Group (PAM)

SUMMARY:
Compare the Effect of Different Physical Programs on the Body Composition of Adult Women and Men With a Total Body Fat Percentage ≥ 30 % at the Beginning of the Test or BMI ≥25

DETAILED DESCRIPTION:
Weight loss by exercise can be frequently deceptive. The focus continues to be centred around total body weight and body mass index (BMI), despite the fact that body fat and fat-free mass are the indicators that represent the greatest risk in the comorbidity associated with obesity. Body weight per se cannot be considered to be reliable; however, its quality can be justified, when measured together with the loss in body fat and the maintenance or increase in fat-free mass.

The purpose of the study is compare the effect of different physical programs (FA) on the body composition (BC) of adult women with a total body fat percentage ≥ 30 % and adult men with a BMI ≥25 at the beginning of the test.

Participants (n=220, women = 110, men = 110) will be recruited through outpatient from private clinics in Cádiz, Andalucía, Spain, as well as through community presentations. Overweight or obese and sedentary women and men will be randomly assigned into three groups according to different levels of AF. 21 of the participants will be assigned to the sedentary control group (METs <2.9), 20 in a group of moderate AF (METs 3-5.9), and 19 will be assigned to the group of intense AF (METs >6).

For 6 months, all of the women shall follow the same diet with an identical distribution of macronutrients. There will be a weekly check up of weight, fat, body water and muscle mass for all of them.

ELIGIBILITY:
Inclusion Criteria:

* Having a body fat percentage >30
* Having a BMI >25
* Being sedentary and
* Have not been submitted to a restrictive diet in the 6 months preceding this study.

Exclusion Criteria:

* Suffered from type 2 diabetes or renal conditions
* Being pregnancy or attempt at pregnancy,
* Being in a maternal lactation period,
* Being underage
* Undergoing antidepressant pharmacological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline BMI. | At baseline (0 years) and followed for 2 years
  Baseline mean BMI values will be measured and compared at 3, 6, 12 and 24 months. BMI will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale.
Changes from baseline Fatty mass. | At baseline (0 years) and followed for 2 years
  Baseline mean Fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Free-fatty mass. | At baseline (0 years) and followed for 2 years
  Baseline mean Free-fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Free-fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Muscular Mass. | At baseline (0 years) and followed for 2 years
  Baseline mean Muscular Mass values will be measured and compared at 3, 6, 12 and 24 months. Muscular Mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Changes from baseline Corporal Water . | At baseline (0 years) and followed for 2 years
  Baseline mean Corporal Water values will be measured and compared at 3, 6, 12 and 24 months. Corporal Water will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Adherence to dietary pattern will be also measured through personal interview | At baseline (0 years) and followed for 2 years
  Participants will be subjected for an intervention based on nutritional (control group) and physical education (two intervention arms) during 24 months. Partial measures will be also taken every week. In the end of the trial, changes in dietary patterns will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.
Adherence to physical activity patterns will be also measured through IPAQ (International Physical Activity Questionnaire). | At baseline (0 years) and followed for 2 years
  Participants will be subjected for an intervention based on nutritional (control group) and physical education (two intervention arms) during 24 months. Partial measures will be also taken every week. In the end of the trial, changes in physical activity will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Hernández-Reyes, Principal Investigator — Universidad de Córdoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez-Reyes A, Camara-Martos F, Molina-Luque R, Romero-Saldana M, Molina-Recio G, Moreno-Rojas R. Changes in body composition with a hypocaloric diet combined with sedentary, moderate and high-intense physical activity: a randomized controlled trial. BMC Womens Health. 2019 Dec 27;19(1):167. doi: 10.1186/s12905-019-0864-5. PMID 31882009